CLINICAL TRIAL: NCT04918459
Title: EUS Guided Cyanoacrylate Injection vs Endoscopic Variceal Band Ligation for Prevention of Rebleeding in Patients With Hepatocellular Carcinoma and Esophageal Variceal Bleeding: a Retrospective Comparative Study
Brief Title: EUS Glue vs Endoscopic Variceal Band Ligation for Prevention of Rebleeding in Patients With HCC and EV Bleeding: a Retrospective Comparative Study
Acronym: EUSgluevsVBL
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Assitant Professor, Chinese University of Hong Kong
Other Study IDs: 2021.221
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: EUS Guided Cyanoacrylate Injection; Endoscopic Variceal Band Ligation; Hepatocelular Carcinoma; Esophageal Variceal Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUS guided cyanoacrylate injection: EUS guided cyanoacrylate injection to prevent EV rebleeding.
- variceal band ligation: variceal band ligation to prevent EV rebleeding.

SUMMARY:
SP by EUS-CYA improves clinical outcomes (eg, EV rebleeding) in patients with HCC and prior EV bleeding when compared with SP by EGD-VBL

DETAILED DESCRIPTION:
Variceal bleeding is a life-threatening complication in patients with portal hypertension and cirrhosis. Rebleeding is common in patients who survive the acute variceal bleeding episode without secondary prophylaxis (SP). Hepatocellular carcinoma (HCC) and portal vein thrombosis (PVT) are associated with recurrent variceal bleeding and worse clinical outcomes. Rebleeding rates of esophageal varices (EV) and gastric varices (GV) remain substantial in HCC patients despite conventional endoscopic treatments.

Lack of SP was associated with a higher rate of rebleeding and mortality in a multicenter study of HCC patients with prior EV bleeding. SP of variceal rebleeding in suitable HCC patients has been suggested in the latest practice guideline of the American Association for the Study of Liver Diseases, but the optimal endoscopic approach for SP in HCC patients has not been well defined. Whether conventional strategies such as variceal band ligation (VBL) or cyanoacrylate (CYA) injection for EV can achieve durable variceal control in HCC patients remains unclear since HCC patients were often excluded from clinical trials. This remains a pertinent issue as recent advances in the treatment of advanced HCC with tyrosine kinase inhibitors (TKI) and immunotherapy means that some patients may achieve reasonable survival and benefit from further variceal management.

Recently, endoscopic ultrasound (EUS) guided variceal interventions by CYA, coiling, or a combination of both have gained clinical attention due to its high clinical success. When compared with conventional endoscopic variceal treatments, EUS guided variceal interventions allow real-time confirmation of intra-variceal delivery of therapy and flow obliteration after treatment. A recent study from our group reported that SP by EUS-CYA reduced rebleeding rate and improved variceal bleeding-free survival in patients with inoperable HCC and variceal bleeding when compared with no SP. However, there has been no dedicated study comparing the clinical outcomes of SP by EUS guided CYA (EUS-CYA) or conventional VBL by esophagogastroduodenoscopy (EGD) in patients with HCC and EV bleeding. Therefore, we propose this retrospective study to compare the clinical outcomes after EUS-CYA or EGD-VBL for SP of EV rebleeding in this often difficult-to-treat patient group with HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive HCC patients with history of EV bleeding who underwent EUS guided cyanoacrylate injection or variceal band ligation by EGD for secondary prophylaxis to prevent EV rebleeding
2. Age > 18 years

Exclusion Criteria:

1. HCC patients with non-variceal upper GI bleeding
2. HCC patients with history of EV bleeding who did not undergo further endoscopy for secondary prophylaxis for EV rebleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC apatients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Death adjusted cumulative incidence of rebleeding at 30-day | 30 days
  Death adjusted cumulative incidence of rebleeding at 30-day

SECONDARY OUTCOMES:
Death adjusted cumulative incidence of rebleeding at 90-day | 90 days
  Death adjusted cumulative incidence of rebleeding at 90-day
Bleeding-free survival at 3 months and 6 months | 6 months
  Bleeding-free survival at 3 months and 6 months
Adverse events related to EUS-CYA or EGD-VBL for secondary prophylaxis | during EUS procedure
  Adverse events related to EUS-CYA or EGD-VBL for secondary prophylaxis
Mortality rate at 6 months | 6 months
  Mortality rate at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tang, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No